CLINICAL TRIAL: NCT07201181
Title: Prenatal Tobacco Exposure Categorized by Maternal Cotinine (Active, Passive, None) and Its Association With Neonatal Metabolic and Physiologic Indices: A Single-Center Prospective Cohort
Brief Title: Maternal Smoking Exposure and Newborn Outcomes: Study Using Urinary Cotinine
Status: Not yet recruiting | Type: Observational
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Berker Okay, MD - Pediatrician (Principal Investigator), Haseki Training and Research Hospital
Other Study IDs: 141-2025
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Tobacco Smoke Pollution; Maternal Exposure During Pregnancy; Infant, Newborn; Carbon Monoxide Poisoning
Keywords: Urinary Cotinine; Prenatal Tobacco Exposure; Maternal Smoking
MeSH Terms: conditions — Carbon Monoxide Poisoning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Maternal Active Smoking (Cotinine-Defined): Mother reports active cigarette smoking during pregnancy and urinary cotinine consistent with active smoking per laboratory cutoffs. Newborn outcomes (cord blood gas incl. pH/base excess/lactate, FCOHb), birthweight, 6-hour blood pressure/vitals, heel-prick TSH, hearing screen, and routine labs are recorded within 24 hours of birth. No experimental intervention is administered.
- Maternal Passive Tobacco Exposure (Secondhand; Cotinine-Defined): Mother denies active smoking but reports secondhand exposure; urinary cotinine detectable yet below active-smoker threshold per laboratory cutoffs. Same neonatal measurements and timing as other cohorts; no experimental intervention.
- No Tobacco Exposure (Reference): Mother denies smoking and secondhand exposure; urinary cotinine negative/undetectable per laboratory cutoffs. Same neonatal measurements collected within routine care; no experimental intervention.

SUMMARY:
Prenatal exposure to tobacco smoke-whether from active maternal smoking or secondhand exposure-has been linked to adverse neonatal adaptation and metabolic stress. This single-center prospective observational cohort will quantify maternal smoking exposure using maternal urinary cotinine around delivery and examine its association with early neonatal physiologic and biochemical outcomes within the first 24 hours of life.

Participants will be pregnant individuals delivering at a tertiary academic hospital and their newborns. After consent, mothers will provide a urine sample for cotinine measurement. Based on pre-specified cotinine thresholds and maternal history, dyads will be classified into three exposure groups: Active smoker, Passive exposure, or No exposure. No experimental intervention is administered; all neonatal assessments are part of routine peripartum care.

Neonatal data collected (per standard practice) will include: umbilical cord blood gas parameters (pH, base excess, lactate) and fetal carboxyhemoglobin (FCOHb); birthweight; vital signs/blood pressure at ~6 hours; routine laboratory indices (e.g., hemogram, lipids such as HDL/LDL where available per unit protocol); heel-prick TSH from the standard newborn screen; and hearing screening result prior to discharge. Additional maternal and perinatal covariates (e.g., age, parity, gestational age, delivery mode, intrapartum events) will be recorded to support adjusted analyses. No extra phlebotomy beyond standard care will be performed; the study leverages existing clinical samples and measurements.

Primary objective is to determine whether higher maternal cotinine-defined exposure is associated with greater metabolic stress at birth (indexed by cord lactate and related gas parameters) and higher FCOHb. Key secondary objectives include evaluating associations with birthweight, early blood pressure, TSH, hearing screen outcomes, and routine laboratory markers. Prespecified subgroup and sensitivity analyses (e.g., by gestational age strata or delivery mode) will be conducted as feasible.

The planned sample includes approximately three cotinine-stratified cohorts recruited consecutively. Statistical analyses will follow a pre-registered plan using multivariable regression to adjust for confounders; ROC analyses may be used to explore cotinine thresholds predictive of adverse neonatal indices. Enrollment is anticipated to start October 13, 2025, with primary data collection completed within 2-3 months of recruitment initiation.

This study will provide pragmatic, prospectively collected evidence on how biochemically verified maternal tobacco exposure relates to immediate neonatal metabolic, cardiovascular, endocrine, and auditory outcomes, using measurements obtainable in routine care.

ELIGIBILITY:
Inclusion Criteria:

* Liveborn neonate delivered at the study hospital, aged 0-72 hours at assessment.
* Routine umbilical cord blood gas available at birth (pH, base excess, lactate).
* Maternal urinary cotinine available around delivery (to classify exposure: active, passive, none).
* Parent/guardian provides informed consent for use of neonatal data obtained from routine care.
* Standard newborn assessments obtainable within 72 hours (e.g., birthweight, ~6-hour vitals/BP, TSH at 24-48 h, hearing screen ≤72 h per unit practice).

Exclusion Criteria:

* Emergent clinical scenarios where any research step could delay urgent care.
* Major congenital anomaly/condition that precludes standard assessments (e.g., cord gas not feasible) per clinician judgment.
* No maternal urine available for cotinine measurement (exposure cannot be defined).
* Prior enrollment of the same neonate (no re-enrollment).

Ages: 0 Minutes to 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Single-center tertiary hospital; consecutively recruited newborns (0-72 h) at birth/discharge. Neonates are stratified by maternal urinary cotinine (Active smoker, Passive exposure, No exposure). Outcomes are sourced exclusively from routine care within 72 h: cord blood gas (pH, BE, lactate) and FCOHb if available; birthweight; ~6-hour blood pressure/vitals; heel-prick TSH (24-48 h); hearing screen (≤72 h); and routine labs (e.g., CBC; HDL/LDL if obtained). No experimental interventions; no extra phlebotomy.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2025-10-13 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Umbilical Cord Blood Lactate | At birth (sample obtained within 10 minutes of delivery; analyzed within routine lab turnaround)
  Cord blood lactate (mmol/L) measured per standard laboratory protocol. Primary analysis compares lactate across cotinine-defined exposure groups (active vs passive vs none) with multivariable adjustment (e.g., gestational age, mode of delivery). No extra blood drawn beyond routine cord sampling.
  Unit of Measure: mmol/L

SECONDARY OUTCOMES:
Umbilical Cord Blood pH | At birth (within 10 minutes)
  Arterial/venous cord blood pH per routine gas analysis; association with maternal cotinine exposure categories.
  Unit of Measure: pH units
Umbilical Cord Blood Base Excess (BE) | At birth (within 10 minutes)
  Base excess from routine cord gas; group comparisons and adjusted models parallel to primary analysis.
  Unit of Measure: mEq/L
Fetal Carboxyhemoglobin (FCOHb) | At birth (same cord sample, routine CO-oximetry if available)
  Percent carboxyhemoglobin from cord blood CO-oximetry; tested for dose-response with maternal urinary cotinine.
  Unit of Measure: percent

REFERENCES:
- [Background] Abraham M, Alramadhan S, Iniguez C, Duijts L, Jaddoe VW, Den Dekker HT, Crozier S, Godfrey KM, Hindmarsh P, Vik T, Jacobsen GW, Hanke W, Sobala W, Devereux G, Turner S. A systematic review of maternal smoking during pregnancy and fetal measurements with meta-analysis. PLoS One. 2017 Feb 23;12(2):e0170946. doi: 10.1371/journal.pone.0170946. eCollection 2017. PMID 28231292
- [Background] Filis P, Hombach-Klonisch S, Ayotte P, Nagrath N, Soffientini U, Klonisch T, O'Shaughnessy P, Fowler PA. Maternal smoking and high BMI disrupt thyroid gland development. BMC Med. 2018 Oct 23;16(1):194. doi: 10.1186/s12916-018-1183-7. PMID 30348172
- [Background] Di HK, Gan Y, Lu K, Wang C, Zhu Y, Meng X, Xia WQ, Xu MZ, Feng J, Tian QF, He Y, Nie ZQ, Liu JA, Song FJ, Lu ZX. Maternal smoking status during pregnancy and low birth weight in offspring: systematic review and meta-analysis of 55 cohort studies published from 1986 to 2020. World J Pediatr. 2022 Mar;18(3):176-185. doi: 10.1007/s12519-021-00501-5. Epub 2022 Jan 28. PMID 35089538
- [Background] Berlin I, Heilbronner C, Georgieu S, Meier C, Spreux-Varoquaux O. Newborns' cord blood plasma cotinine concentrations are similar to that of their delivering smoking mothers. Drug Alcohol Depend. 2010 Mar 1;107(2-3):250-2. doi: 10.1016/j.drugalcdep.2009.10.008. Epub 2009 Nov 24. PMID 19939584
- [Background] Hayde M, Bernaschek G, Stevenson DK, Knight GJ, Haddow JE, Widness JA. Antepartum fetal and maternal carboxyhemoglobin and cotinine levels among cigarette smokers. Acta Paediatr. 1999 Mar;88(3):327-31. doi: 10.1080/08035259950170123. PMID 10229047
- [Background] Wang X, Tager IB, Van Vunakis H, Speizer FE, Hanrahan JP. Maternal smoking during pregnancy, urine cotinine concentrations, and birth outcomes. A prospective cohort study. Int J Epidemiol. 1997 Oct;26(5):978-88. doi: 10.1093/ije/26.5.978. PMID 9363518